CLINICAL TRIAL: NCT02774655
Title: New Health Devices to Improve Adherence to Physical Activity in Overweight Inactive Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2015/1750
Record Dates: First submitted 2016-05-13; First posted 2016-05-17 (Estimated); Last update posted 2017-09-25 (Actual); Status verified 2017-09

CONDITIONS: Cardiovascular Diseases; Obesity
Keywords: healthy volunteers; patient compliance; exercise; motivation
MeSH Terms: conditions — Cardiovascular Diseases; Obesity; Patient Compliance; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PAI APP (Experimental): personal activity index application
  Interventions: Device: Pai APP
- FitBit APP (Active Comparator)
  Interventions: Device: FitBit APP

INTERVENTIONS:
Device: Pai APP — prescribed 100 PAI weekly
  Other Names: personal activity Intelligence (PAI) application; Mio Fuse wristband
  Arms: PAI APP
Device: FitBit APP — prescribed 10000 steps daily
  Other Names: FitBit zip step counter
  Arms: FitBit APP

SUMMARY:
The purpose of this study is to test in overweight and inactive adults whether the new PAI eHealh APP leads to better adherence to a physical activity regimen than the wearable step counter App from the market leader FitBit, and to evaluate if improved adherence will be reflected in a better cardiovascular profile in this group.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index > 25
* self reported exercise one time or less per week

Exclusion Criteria:

* inability to use a SmartPhone
* illness or disabilities that preclude or hinder completion of the study
* cancer that makes participation impossible or exercise contraindicated (considered individually, in consultation with physician)
* test results indicating that study participation is unsafe
* participation in other studies conflicting with participation in this study
* symptomatic valvular, hypertrophic cardiomyopathy, unstable angina, primary pulmonary hypertension, uncontrolled hypertension, heart failure or sever arrhythmia
* diagnosed dementia
* chronic communicable infectious diseases
* Bariatric surgery
* Medication for thyroid disease, diabetes, blood pressure or lipid lowering medication

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
The proportion of the participants obtaining 80 % or more of the prescribed physical activity for one year | 1 year
  Prescribed 100 PAI weekly (PAI app group), or 10 000 steps daily (step counter app)

SECONDARY OUTCOMES:
Cardiorespiratory fitness | 1 year
  Peak oxygen uptake assessed by Jaeger oxycon pro; Erich Jaeger GmbH, Hoechberg, Germany
Cardiorespiratory fitness | 16 weeks
  Peak oxygen uptake assessed by Jaeger oxycon pro; Erich Jaeger GmbH, Hoechberg, Germany
Resting blood pressure | 16 weeks
  Left upper arm, right upper arm, orthostatic hypotension
Resting blood pressure | 1 year
  Left upper arm, right upper arm, orthostatic hypotension
Resting heart rate | 16 weeks
Resting heart rate | 1 year
Body mass index | 16 weeks
  Height, weight
Body mass index | 1 year
  Height, weight
Waist line | 16 weeks
  in centimeters
Waist line | 1 year
  in centimeters
Body composition | 16 weeks
  body composition measured by bioelectrical impedance (InBody 720, BIOSPACE, Seoul, Korea)
Body composition | 1 year
  body composition measured by bioelectrical impedance (InBody 720, BIOSPACE, Seoul, Korea)
Activity questionnaire | 16 weeks
  HUNT-1 questionnaire 2 "exercise"
Activity questionnaire | 1 year
  HUNT-1 questionnaire 2 "exercise"
glucose concentration in blood | 16 weeks
glucose concentration in blood | 1 year
glycosylated haemoglobin (HbA1c) concentration in blood | 16 weeks
glycosylated haemoglobin (HbA1c) concentration in blood | 1 year
c-peptide concentration in blood | 16 weeks
c-peptide concentration in blood | 1 year
concentration of triglycerides in blood serum | 16 weeks
concentration of triglycerides in blood serum | 1 year
concentration of total cholesterol in blood | 16 weeks
concentration of total cholesterol in blood | 1 year
concentration of low density lipid (LDL) cholesterol in blood | 16 weeks
concentration of low density lipid (LDL) cholesterol in blood | 1 year
concentration of high density lipid (HDL) cholesterol in blood | 16 weeks
concentration of high density lipid (HDL) cholesterol in blood | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Ulrik Wisløff, prof, Study Director — Norwegian University of Science and Technology
Locations (1):
- Institutt for sirkulasjon og bildediagnostikk, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: Undecided